CLINICAL TRIAL: NCT02048748
Title: Congestive Heart Failure Home Telemonitoring : A Home Telemonitoring Service for Chronic Heart Failure Patients on Trial
Brief Title: Congestive Heart Failure Home Telemonitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was ended before any patients were enrolled. Department of Clinical Research, August 2020.
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UNN-NST-TeleCHF-01
Record Dates: First submitted 2013-10-30; First posted 2014-01-29 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2014-01

CONDITIONS: Heart Failure; Blood Pressure; Body Weight
Keywords: Home Care Services; Telemedicine
MeSH Terms: conditions — Heart Failure; Body Weight | interventions — Weights and Measures; Sphygmomanometers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental): Device: Weight and blood pressure device Device: Home telemonitoring device
  Interventions: Device: Weight and blood pressure device; Device: Home telemonitoring device
- Control (No Intervention): Usual care

INTERVENTIONS:
Device: Weight and blood pressure device — Weight and blood pressure device integrated in a home telemonitoring kit. The weight scale is Withings The Smart Bodyscale. The blood pressure device is MEDISANA iHealth BP3.
  Arms: Telemonitoring
Device: Home telemonitoring device — An iPad 2 WiFi 16GB (Model A1395) tablet integrating the telemonitoring kit.
  Arms: Telemonitoring

SUMMARY:
Remote monitoring of chronic heart failure can reduce deaths and hospitalisations, and may provide benefits on health care costs and quality of life. Currently there is limited use of remote monitoring for heart failure in Norway. The funding streams and the structure of the norwegian health service is different from other countries that have tried remote monitoring and therefore it is important to examine the utility of such services in Norway. The study is a randomised controlled trial that will allow participants in the intervention group to use a wireless weight scale and blood pressure monitor device that will send automatically the measurements electronically and securely to the Heart Failure Outpatient Clinic of the hospital.

DETAILED DESCRIPTION:
Providing patients with chronic heart failure (CHF) access to remote monitoring, for example by telephone or telemonitoring using wireless technology, reduces deaths and hospitalisations and may provide benefits on health care costs and quality of life. Remote monitoring of patients can reduce pressure on resources, particularly for conditions like chronic heart failure, which exert a large burden on health services. These are conclusions of a Cochrane Systematic Review.

In Norway the costs for treatment of chronic heart failure are vast, both concerning hospital treatment, daily use of medication over years, and loss of quality of life for patients and their family caregivers. Generally there is little knowledge about what is gained for the billions used. In Norway no telemonitoring services are established and hence no investigations have yet been published. Thus it seems that current evidence of effectiveness and quality is insufficient to recommend usage. The structure and funding streams in Norwegian health services are different from other countries and the conventional services that the intervention has been compared to in previous studies, are most likely heterogeneous. It is thus important to investigate Norwegian conditions.

Advanced telemonitoring technology with electronic transfer of physiological data such as blood pressure and weight is currently being used in research and established routine services in several countries in Europe, amongst them the Netherlands, Germany and the United Kingdom.

The proposed project intends to introduce such a strategy as an avenue for exploring promising new services that would not otherwise be available in Norway. The service consists of daily monitoring the patients' weight and blood pressure directly from their home; automatically and securely transmit the values to a server at UNN; and monitor the values by a trained nurse at the Heart polyclinic.

The primary objective of this study is thus to explore whether, as compared to current care from the heart polyclinic, the introduction of home telemonitoring will reduce hospital readmissions and will, in addition, be cost-effective. This is in line with the recent directions of European telemonitoring programmes for patients with chronic heart failure. This result may define if the telemonitoring of heart failure patients is feasible for Norway or not at all.

Identifying successful innovations to be introduced into the Norwegian health care services is a condition for more cost effectiveness and better treatment quality.

ELIGIBILITY:
Inclusion Criteria:

* the presence of CHF signs and symptoms such as dyspnoea and peripheral or pulmonary oedema requiring diuretic administration (New York Heart Association [NYHA] functional class II-IV); and
* ejection fraction (EF) under 40% combined or not with a left ventricular filling pattern supporting the presence of diastolic dysfunction, according to the American College of Cardiology/American Heart Association Guidelines for chronic heart failure.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
CHF related hospital readmissions | 12 months

SECONDARY OUTCOMES:
Length of stay | 12 months
  Length of stay per hospitalisation
Quality of Life MLwHF | 6 months, 12 months
Challenges and opportunities | 12 months
  Qualitative analysis of conditions for identified best practices resulting from the intervention, and possible to be developed. Interview with patients and health professionals. Thematic analysis of transcribed interviews. Identification of themes related to best practices and challenges.
Additional costs/savings resulting from the service | 12 months
  Additional costs/savings resulting from the service defined as the difference in the costs of medical care during the study, identified through a cost analysis, between the intervention and control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Artur Serrano, PHD, Principal Investigator — Norwegian Centre for Integrated Care and Telemedicine
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- See also: Norwegian Centre for Integrated Care and Telemedicine — http://www.telemed.no